CLINICAL TRIAL: NCT04521127
Title: Comparison of Dry Needling and Kinesio Taping Methods in the Treatment of Myofascial Pain Syndrome
Brief Title: Dry Needling and Kinesio Taping in the Treatment of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physical Med-1
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Myofascial Pain Syndrome of Neck
Keywords: Taping; Pain; Trigger Point; Dry needling
MeSH Terms: conditions — Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Three groups with a conventional therapy control group.
Who Masked: Outcomes Assessor
Masking Description: Patients will be aware of group distribution due to the nature of the taping and DN procedures. Therefore, the only outcome assessor will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Taping Group (Active Comparator): Kinesio taping will be applied to trapezius muscle
  Interventions: Other: Kinesio Taping
- Dry needling Group (Active Comparator): Dry needling will be applied to trigger point on trapezius muscle
  Interventions: Other: Dry needling
- Control Group (No Intervention): Control group will not receive any additional intervention

INTERVENTIONS:
Other: Kinesio Taping — Taping will be performed on sitting position with contralateral lateral flexion and flexion of the neck, using muscle technique with I strip and stretching the head at the maximum level in order to benefit from the muscle release effect. Kinesio tape was applied directly on muscle with 0% stretching.
  Arms: Kinesio Taping Group
Other: Dry needling — The trigger point on the taut band will be held with the thumb and forefinger from below and above. In the needling technique, a 0.25 * 25-mm with nickel handle, disposable sterile steel acupuncture needle will be used. The needle tip will be inserted perpendicularly into the subcutaneous tissue and inserted into the muscle until the trigger point in the taut band was found. The same point will be pinned 8-10 times with fast needle movements inside and out. Then the needle tip will pulled back so that it did not come out of the skin, and the bottom, top and sides of the first entered point were also pinned. This procedure was applied to all trigger points in the trapeze muscle.
  Arms: Dry needling Group

SUMMARY:
The aim of this study is to compare the effectiveness of kinesio tape and dry needling in the treatment of myofascial pain syndrome of the trapezius muscle.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a common problem with manifesting itself such as trigger points, taut bands, range of motion limitations and pain. One of the most common place for MPS is neck region and trapezius muscle is the common cause of these symptoms and 9 different trigger point location has been identified on trapezius muscle. Myofascial trigger points, characterized by hypersensitive nodules, can be palpated in stretched bands in the affected muscles. In order to eliminate trigger points fascial releasing, dry needling, kinesio taping and other physical therapy applications can be used.

Although there are several studies investigating the effectiveness of Kinesio taping (KT) and Dry needling(DN) methods in MPS, it is controversial which one is superior to others.

The aim of this study is to compare the effects of exercise, KT, and DN methods on pain and disability in the treatment of upper trapezoidal muscle MPS.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosis with MPS and having active myofascial trigger points on trapezius muscle

Exclusion Criteria:

* Fibromyalgia
* a history of myofascial trigger point injection
* acute trauma
* inflammatory joint or muscle disease
* infection or malignancy on cervical region
* neurological disorders
* cervical radiculopathy or myelopathy
* inadequate cooperation for the treatment
* a history of neck surgery or spinal degeneration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) Measurement | two weeks
  Pain pressure threshold (PPT). was assessed with an analogue algometry (Baseline, FEl Inc. White Plains, NY,USA) with 1 cm2 rubber tip was used to measure the pain pressure threshold. Algometer perpendicularly placed over spinous process of T1 on prone position and pressure progressively increased 1 kg/s until patients verbally reported pain under the tip of algometer or referring pain. Measurement repeated three times and average score recorded.

SECONDARY OUTCOMES:
Visual analog scale | two weeks
  The patient was asked to mark the severity of his or her pain with active motion on a horizontal line 100 millimeters in length. The intensity of the pain was calculated by measuring the area in which the individual marked between 0 (no pain) and 10 (the most severe pain I felt in my life).
Neck Disability Index | two weeks
  Perceived disability of patients was assessed with 10-item item Neck Disability Index (NDI),which a modified from Oswestry Low Back Pain Disability Index to assess with a score range of 0 to 50.
Global Perceived Effect Scale | two weeks
  Change in the perception of the symptoms after the treatment was measured by a Global Perceived Effect Scale. Patients were asked to rate change between 1 completely recovered, 4 unchanged, 7 vastly worse on a horizontal likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Fatih Yaşar, MD, Principal Investigator — Bolu Abant Izzet Baylsa University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No